CLINICAL TRIAL: NCT05057624
Title: Gaze-Contingent Music Reward Treatment (GC-MRT) for PTSD
Brief Title: Gaze-Contingent Music Reward Treatment for PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a lack of funding, this study was not initiated.
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Principal Investigator, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: # 7960
Record Dates: First submitted 2021-08-31; First posted 2021-09-27 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- non-GC-MRT (Placebo Comparator): Placebo- music will play at all times during the trials.
  Interventions: Other: Placebo GC-MRT
- GC-MRT (Active Comparator): Music will only play when participants view angry faces and will stop when they look at neutral faces.
  Interventions: Other: GC-MRT
- GC-MRT-exp (Experimental): Music will only play when participants look at neutral faces and will stop when they view angry faces.
  Interventions: Other: Exposure

INTERVENTIONS:
Other: Placebo GC-MRT — Participants will hear music continuously throughout the trials, without regard to the faces they look at.
  Other Names: Control
  Arms: non-GC-MRT
Other: GC-MRT — Participants will hear music as a reward for looking at neutral faces and the music will stop when they focus on angry faces.
  Arms: GC-MRT
Other: Exposure — Participants will hear music of their choice when they focus on angry faces, and when they look at neutral faces the music will stop.
  Other Names: GC-MRT-Exp
  Arms: GC-MRT-exp

SUMMARY:
The present study is a double-blind trial that seeks to examine the feasibility, acceptability, and efficacy of a recently developed eye-tracking-based, gaze-contingent music reward therapy (GC-MRT) in individuals with posttraumatic stress disorder (PTSD).

The specific aims of this study are to: (1) examine the efficacy of GC-MRT in PTSD; and (2) elucidate its underpinnings (i.e. attention control, reward processes, and exposure via counter-conditioning).

The investigators hypothesize that:

1. GC-MRT will produce greater reductions in symptoms compared to PC at post-treatment and follow-up (diverting attention away from threat).
2. GC-MRT-exp will produce greater reductions in symptoms compared to PC at post-treatment follow-up (exposure via counter-conditioning by rewarding threat stimuli).
3. Exploratory analysis will compare the reductions in symptoms of GC-MRT compared to GC-MRT-exp at post-treatment follow-up.

DETAILED DESCRIPTION:
GC-MRT is designed to shift participants' attention away from threat and toward neutral stimuli by introducing a contingency between viewing patterns and music pre-chosen by participants. Participants view matrices of faces with neutral and angry expressions. Viewing the neutral faces triggers music the participant previously requested, and viewing the angry faces turns the music off. The researchers will compare this condition (GC- MRT) to two additional conditions. In the "exposure" condition (GC-MRT-exp) the investigators will reverse the music contingency such that viewing the angry faces triggers the music while viewing the neutral faces turns the music off. In the placebo control (PC) condition, music plays continuously.

The goal of this study is to: (1) examine the efficacy of GC-MRT in PTSD; and (2) elucidate its underpinnings (i.e. attention control, reward processes, and exposure via counter-conditioning).

Attention control is the ability to shift attention deliberately based on goal-directed behavior. Accordingly, deficits in attention control can result in volatile shifts in attention leading to increase attention allocation to threat in the environment.

Reward functioning is the ability to seek out and enjoy stimuli of positive motivational valence, and is considered a crucial driving force of behavior, guiding the organism towards positive and rewarding experiences, ranging from food and gender to money, music, and positive social interactions.

Allocating visual attention to rewarding stimuli is considered a reward-related attentional feature.

Counter-conditioning is an alternative to exposure therapy involving pairing of the feared stimulus with an appetitive/positive outcome (i.e., increasing the rewarding/positive value of the feared stimulus), in which repeated trials are supposed to reduce the fear response, and replace it by an appetitive response. Indeed, studies have shown counter-conditioning to be more effective at reducing fear than traditional exposure therapy.

The investigators hypothesize that:

1. GC-MRT will produce greater reductions in symptoms compared to PC at post-treatment and follow-up (diverting attention away from threat).
2. GC-MRT-exp will produce greater reductions in symptoms compared to PC at post-treatment follow-up (exposure via counter-conditioning by rewarding threat stimuli).
3. Exploratory analysis will compare the reductions in symptoms of GC-MRT compared to GC-MRT-exp at post-treatment follow-up.

Subject population: Seventy-five subjects with PTSD will participate in this study.

Methods: The sample (N = 75) will be randomized equally into three groups. Group 1 will receive a 4-week (8 sessions) course of GC-MRT where music will play only when viewing neutral faces, Group 2 will receive a 4-week (8 sessions) course of GC-MRT-exp where music will play only when viewing angry faces, and Group 3 will receive a 4-week (8-sessions) course of non-GC-MRT (i.e. placebo control; PC) where music will play throughout the trials.

*The pictures of the faces used in the intervention will include 50% male and 50% female. Race-wise they are homogenous. Varying the different faces by race is not feasible as these faces were chosen from an established picture data-base (i.e., the Karolinska Directed Emotional Faces database; KDEF) based on the affective ratings of each face. Importantly, this composition of faces is similar to one used in an attention assessment task for which our pilot data shows significant group differences in dwell time, which is the attentional target of the intervention. Hence, we do not expect this to affect the results.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 80
* Current DSM-5 diagnosis of PTSD
* CAPS-V score greater than or equal to 25
* Fluent in English and willing to give informed written consent and participate responsibly in the protocol.
* Normal or corrected-to-normal vision
* Mini Mental Status Exam score greater than or equal to 24.

Exclusion Criteria:

* History of psychiatric diagnosis of psychotic episode, psychotic disorder, schizophrenia, schizoaffective disorder
* Current severe depression determined by a a) score greater than 25 on the Hamilton Rating Scale for Depression (HAM-D-17) and evaluation and b)clinical assessment
* Suicidal ideation or behavior
* Current or past diagnosis of obsessive compulsive disorder, bipolar disorder, epilepsy, or brain injury as determined by a Structured Clinical Interview for DSM-5 (SCID-5) interview
* Current or past organic mental disorder, seizure disorder, epilepsy or brain injury as determined by a clinical evaluation
* Diagnosis of probable Alzheimer's disease, Vascular Dementia, or Parkinson's Disease, as determined by a clinical evaluation and Mini Mental Status Exam (MMSE)
* Current unstable or untreated medical illness
* Drug or alcohol misuse- severe alcohol/cannabis disorder or any other substance use disorder except nicotine.
* Recurrent psychotropic medication change or initiation within the last 3 months
* Initiation of psychotherapy within the last 3 months
* Current or past Attention Deficit Hyperactivity Disorder (ADHD) diagnosis
* Chronic pain that may affect sitting down and still for approximately 30 minutes
* Current cognitive impairments as a result of a traumatic brain injury, as determined by a clinical evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-09-14 (Estimated); Study Completion 2025-03-14 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms over time | Baseline, at 5 weeks, posttreatment at 10 weeks, follow up at 3 months from last session
  Reduction in symptoms as measured by the Clinician Administered PTSD Scale (Caps-5: ranging from 0-80 ). from pre- to post-treatment. Lower scores mean better outcome
Change in depressive symptoms over time | Baseline, at 5 weeks, posttreatment at 10 weeks, follow up at 3 months from last session
  Change in symptoms as measured by the Hamilton Depression Rating Scale (HDRS-17; range 0-52) from pre- to post-treatment.
Change in anxiety symptoms over time | Baseline, at 5 weeks, posttreatment at 10 weeks, follow up at 3 months from last session
  Change in symptoms as measured by the Hamilton Anxiety Rating Scale (HAM-A); range 0-56) from pre- to post-treatment.
Changes in illness severity and improvement over time | Baseline, at 5 weeks, posttreatment at 10 weeks, follow up at 3 months from last session
  Reduction in overall symptoms as measured by the Clinical Global Impressions scale (illness severity rated 0 to 7, with higher scores indicating more severe illness; improvement rated 0 to 7, with higher scores indicating less improvement.)
Change in the severity of PTSD symptoms over time. | Baseline, at 5 weeks, posttreatment at 10 weeks, follow up at 3 months from last session
  Assesses for change in individual symptoms of PTSD and PTSD severity as measured by the Posttraumatic Stress Disorder Checklist (PCL-5). The severity of 20 PTSD symptoms is rated from 0 to 4, with higher numbers indicative of greater severity (score range of 0 to 80.)
Changes in suicidal ideation and depressive symptoms over time. | each treatment session (weeks 2-10)
  Assessment and monitoring of depressive symptoms and suicidal ideation, as measured through the Beck Depression Inventory-II (BDI-II). Scores range from 0 to 63, with higher scores reflecting more severe depression.
Change in the ability to experience pleasure over time. | Baseline, at 5 weeks (midpoint), posttreatment at 10 weeks, follow up at 3 months from last session
  Change in anhedonia from pre- to post-treatment assessment will be assessed using the The Snaith-Hamilton Pleasure Scale (SHAPS: score range: 0-14, higher scores indicate less ability to experience pleasure).
Change in the ability to feel social pleasure over time | Baseline, at 5 weeks (midpoint), posttreatment at 10 weeks, follow up at 3 months from last session
  Change in anhedonia from pre- to post-treatment assessment will be assessed using the the Revised Social Anhedonia Scale (SHAPS: score range: 0-14, higher scores indicate less ability to experience pleasure).
Change in people's experiences of music as a reward over time. | Baseline, at 5 weeks (midpoint), posttreatment at 10 weeks, follow up at 3 months from last session
  Change in people's experiences of music as a reward and their relationship to music, as measured by the Barcelona Music Reward Questionnaire (BMRQ score range: 40-60, with higher scores indicate greater experiences of music as a reward)

IPD SHARING:
Plan to Share IPD: No